CLINICAL TRIAL: NCT04171310
Title: An Open-label Study of Excretion Balance and Pharmacokinetics Following a Single Oral Dose of [14C]-SAR442168 (Not More Than 3.7 MBq) in Healthy Male Subjects
Brief Title: Study of Excretion Balance and Pharmacokinetics of [14C]-SAR442168 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEX16018; 2019-001069-33 (EudraCT Number); U1111-1223-4541 (Other: UTN)
Record Dates: First submitted 2019-11-19; First posted 2019-11-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAR442168 (Experimental): Single oral dose of SAR442168 (as a nonsalified compound) containing (NMT) 3.7 MBq of [14C]-SAR442168
  Interventions: Drug: SAR442168

INTERVENTIONS:
Drug: SAR442168 — Pharmaceutical form:oral solution Route of administration: Oral

SUMMARY:
Primary Objective:

To determine the excretion balance and systemic exposure of radioactivity after oral administration of [14C]-SAR442168.

To determine the pharmacokinetics of SAR442168 and its contribution to the overall exposure of radioactivity.

To collect samples in order to determine the metabolic pathways of SAR442168 and identify the chemical structures and main excretion route of the main metabolites (samples will be analyzed according to metabolic analysis plan and results will be documented in a separate report).

Secondary Objective:

To assess the clinical and biological tolerability of an oral solution of SAR442168.

DETAILED DESCRIPTION:
Total study duration is 3 to 10 weeks, including a screening period of 27 days, treatment period of up to 15 days and a follow-up and end of study of up to 4 weeks.

ELIGIBILITY:
Inclusion criteria :

Healthy male subjects 30 to 65 years of age. Body Mass Index 18 up to 32 kg/m2, inclusive. Signed informed consent. Subjects must agree to the use of an adequate method of contraception for up to 3 months after discharge from the clinical unit

Exclusion criteria:

Radiation exposure exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last five years (including diagnostic X-rays and other medical exposures).

Occupationally exposure to radiation (as defined in the Ionizing Radiations Regulations 2017).

Irregular bowel habits (more than 3 bowel movements/day or less than 1 every 2 days) .

Social habits: smoking, alcohol abuse, drug abuse etc.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose excreted in urine and feces | Day 1 to Day 43
  Fractional and cumulative percentage of radioactive dose excreted in urine and feces of [14C]-SAR442168

SECONDARY OUTCOMES:
Number of subjects with Adverse events | From Day -1 to 43
  Adverse events, spontaneously reported by the subject or observed by the Investigator
Blood/plasma radioactivity ratio | Day 1 up to Day 43
  Blood/plasma radioactivity ratio for Cmax
Blood/plasma radioactivity ratio | Day 1 up to Day 43
  Blood/plasma radioactivity ratio for AUC
Plasma SAR442168 /radioactivity ratio | Day 1 up to Day 43
  Plasma SAR442168 /radioactivity ratio for Cmax
Plasma SAR442168 /radioactivity ratio | Day 1 up to Day 43
  Plasma SAR442168 /radioactivity ratio for AUC

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 8260001, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BEX16018 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25222&tenant=MT_SNY_9011